CLINICAL TRIAL: NCT00885625
Title: 1-Year Longitudinal Follow-up Study of Serologic Responses to 7-valent Pneumococcal Conjugated Vaccination and Opsonophagocytic Activities for Streptococcus Pneumoniae Among Patients With Human Immunodeficiency Virus Infection
Brief Title: 7-valent Pneumococcal Conjugated Vaccination
Acronym: PCV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Hung Chien-Ching, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200805005M
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2010-07-15 (Estimated); Status verified 2010-06

CONDITIONS: Invasive Pneumococcal Disease
Keywords: invasive pneumococcal disease; pneumococcal conjugated vaccine
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: 7-valent pneumococcal conjugated vaccine — 7-valent pneumococcal conjugated vaccine is given twice with 4 weeks apart
  Other Names: Prevenar (Wyeth)

SUMMARY:
Hypothesis: the efficacy of 2 doses 7-valent PCV is equivalent to 1 dose 7-valent PCV.

DETAILED DESCRIPTION:
Background:

Patients with human immunodeficiency virus (HIV) infection have higher incidence and recurrence rates of pneumonia and bacteremia caused by Streptococcus pneumoniae compared with the persons without HIV infection. Before the introduction of highly active antiretroviral therapy (HAART), the rate of invasive pneumococcal bacteremia was 100-fold greater in HIV-infected patients compared to HIV-negative controls. Since the introduction of HAART in 1996, the incidences of several AIDS-related opportunistic infections have significantly declined. However, the incidence of invasive pneumococcal disease in HIV-infected patients who received HAART is still 35~60-fold higher than non-HIV infected adults. The pathogenesis of invasive pneumococcal disease may be related to decrease of IL-8 level. By multivariate analysis, the major risk factors for pneumococcal bacteremia in HIV-infected patients include age, close exposure to children, associated comorbidity, smoking, alcohol abuse, injecting drug use, prior hospitalization, and CD4 count lower than 100 cells/ul; and the protective factors include HAART use and pneumococcal vaccination.

The 23-valent pneumococcal polysaccharide vaccine (PPV) is recommended for HIV-infected adolescents and adults who have CD4 lymphocytes count >/= 200 cells/ul and is optional for persons with a CD4 lymphocytes count <200 cells/ul. Revaccination one time should also be considered if the initial vaccination was given when the CD4 count was <200 cells/ul and if the CD4 count has increased to >200 cells/ul as a result of HAART. In the following years, there were several studies which had demonstrated that 23-valent PPV vaccination was associated with decreased risk of invasive pneumococcal disease. However, HIV-infected patients who do not have HAART therapy have significantly lower magnitude of antibody responses to 23-valent PPV than those receiving HAART and HIV-uninfected persons, and antibodies titers among HIV-infected patients seem to be associated with CD4 count. In addition, though the rates of decline of mean antibody concentrations in HIV-infected patients and in non-HIV-infected individuals were similar during 5 years after vaccination, as a consequence of lower postvaccination antibody concentration in HIV-infected patients, most of the HIV-infected patients have antibody concentrations below protection level within 3 years after vaccination. The impaired immune response to PPV may be due to PPV is T-lymphocyte-independent type 2 antigens (TI-2 antigens) instead of T-lymphocyte-independent type 1 antigens (TI-1 antigens). The response to TI-2 antigens is dependent on the number and function of T lymphocytes for the induction of an antibody response. Once T-lymphocyte's function is impaired, subsequent antibody response is also compromised. Therefore, the long-lasting immunity of PPV seems limited in HIV-infected patients.

The US Food and Drug Administration approved a 7-valent conjugated pneumococcal vaccine (PCV) in 2000. It contains seven S. pneumoniae polysaccharides combined with a carrier protein which is non-toxic mutant diphtheria toxin. With this combination, it can induce a T-cell dependent immune response and memory T and B cells and enhances better secondary antibody response after contact with the pathogen or revaccination. Several studies have demonstrated that 7-valent PCV-primed patients have higher antibody responses that also induce better opsonophagocytic activity in old or immunocompromised patients such as chronic lymphocytic leukemia, liver transplantation, or allogeneic stem cell transplantation. In HIV-infected patients, the efficacy of 7-valent PCV is also associated with CD4 count but the antibody response and opsonophagocytic activity are still better than those induced by PPV vaccination. However, the 7-valent PCV vaccination schedule and the necessity of booster vaccination are still unknown. In addition, long-term immunity to 7-valent PCV and the correlation with CD4 count are also under investigation.

The goal of our study is to compare the quantitative and functional antibody responses to 1-dose 7-valent PCV and 2-doses 7-valent PCV in HIV-infected patients, and also to compare these responses in HIV-infected patients with different categories of CD4 counts.

Materials and Methods:

Study population

350 HIV-infected adults will be recruited from infectious diseases clinics at National Taiwan University Hospital. Persons aged 18 years or greater who have HIV infection documented by enzyme-linked immunosorbent assay (ELISA) and Western Blot testing are eligible. Persons with the following criteria are excluded: immunization with PPV within the past 5 years; current pregnancy, use of another investigational drug within past 4 weeks; or use of intravenous immunoglobulin within last 3 months, or any other vaccination within the past 2 months. Persons with CD4 counts less than 100 cells/ul or under highly active antiretroviral therapy (HAART) are not excluded.

Based on the CD4+ lymphocyte count within 3 months of pneumococcal vaccination, vaccinees are randomly selected, and three categories of patients are defined:

* Group 1: patients with CD4+<200 cells/ul;
* Group 2: patients with CD4+ 200-350 cells/ul and group 3 with CD4+>350 cells/ul.

After receipt of 7-valent PCV, patients continue their routine follow-up at the outpatient clinics for antiretroviral therapy and related HIV care.

Plasma HIV RNA load is quantified using the Cobas Amplicor HIV-1 Monitor test (Cobas Amplicor version 1.5, Roche Diagnostics Corporation, IN) with a lower detection limit of 40 copies/mL, and CD4+ lymphocyte count is determined using FACFlow (BD FACS Calibur, Becton Dickinson, CA). The CD4+ lymphocyte counts and plasma HIV RNA load are monitored every 3 months.

HAART is defined as the combination of at least 3 antiretroviral agents containing two nucleoside reverse transcriptase inhibitors (NRTIs) plus protease inhibitors (PIs) or one non-nucleoside reverse transcriptase inhibitors (NNRTI); or triple NRTIs.

Vaccine administration

Hepavalent conjugate pneumococcal vaccine (Wyeth-Lederle) contain 2μg of capsular polysaccharide from each of six serotypes (4, 9V, 14, 18C, 19F, and 23F) and 4ug of capsular polysaccharide from serotype 6B covalently linked to a total of 20~25 ug of CRM197, a non-toxic mutant diphtheria toxin. After receipt of a single 0.5 ml injection of 7-valent conjugated pneumococcal vaccine, all patients are prospectively followed for 48 weeks. Sequential blood specimens are collected while the patients returned for routine examinations for plasma HIV RNA load and CD4+ lymphocyte count every 3-6 months. The blood specimens are stored at -70 degrees Celsius until determinations of anti-capsular antibody titers are performed. The study is approved by the Institutional Review Board of the hospital, and every patient gives written informed consent.

All patients are sequentially enrolled into two-phase study according to vaccination doses: group 1: two doses of PCV with 4 weeks apart; group 2: one dose PCV. Vaccine will be administrated by study nurses via intramuscular deltoid injections.

Adverse events Subjects will be given a questionnaire to record any adverse event since vaccination for 7 days. They are also advised to call the study nurses for severe side effects. Severe adverse reactions will be ascertained by interview with the subjects by telephone and hospitalization was suggested.

Specimen collection and determinations of anti-capsular antibody titers Blood will be drawn at 0, 4, 12, 24, 36, and 48 weeks and are separated from clotted blood samples by centrifugation and stored at -70 degrees Celsius. The determinations of anti-capsular antibody levels among serially collected blood specimens from each enrolled patient are carried out with ELISA by following the methods described previously with minor modifications.

Briefly, 1 mL of serum is mixed with 10 mg of CWPS (cell wall polysaccharide) and incubated at room temperature on a rocking platform for 30 min. Sera from patients with AIDS who have no antibody to S. pneumoniae serotypes 14, 19F, 23F, or 6B capsules and <1 ug of antibody to CWPS per mL will be used as negative controls. Capsular polysaccharides from S. pneumoniae serotypes 14, 19F, 23F, or 6B are obtained from the American Type Culture Collection (ATCC). These capsular polysaccharides are suspended in phosphate-buffered saline (PBS, pH7.4) at concentration of 10 ug/mL and used directly to coat wells by incubation at 4 degrees Celsius overnight. After washing, blocking is done with PBS containing 1% of bovine serum albumin at 4 degrees Celsius overnight. Duplicate samples of sera are studied in 2-fold serial dilutions, a laboratory reference standard for each serotype that contained known amount of IgG reactive with specific capsular polysaccharide is included in each plate as a positive control. Following washing, this first antibody incubation is performed at 37 degrees Celsius for 2h. After thorough washing of unbounded antibodies to wells, Horseradish Peroxidase (HRP)-conjugated goat antibody to human IgG (ZYMED LABORATORIES INC, South San Francisco, CA) at 1: 2,000 dilution is used to detect IgG, and the reaction is developed 10 min at dark by addition of K-blue substrate (Neogen Corporation, Lexington, Ky., USA), followed by adding 1N sulfuric acid to stop the reaction. All washings between each incubation were done with PBS buffer containing 0.05% Tween 20. Optical density is read in an ELISA reader (SpectraMAX 340, Molecular Devices, Sunnyvale, CA) at a wavelength of 450 nm, with subtraction of optical density of the appropriate blank.

Significant antibody responses are defined as a 2-fold or greater increase of antibody levels following vaccination compared to those at baseline (responders). The laboratory staff who performed the determinations of antibody responses is blinded to the identity and clinical characteristics of the patients, vaccination status, and whether HAART is initiated.

Opsonophagocytic assay (OPK assay)

OPK titer against S. pneumoniae will be measured as described with minor modification. Briefly, the differentiated HL-60 cells are used at an effector/target cell ratio of 400/1. 20 ml of 2-fold serially diluted, 56 degrees Celsius heat inactivated, serum sample is aliquoted into each well of 96-well microtiter plate. 20 ml of S. pneumoniae bacterial suspension (~103 cfu/well) is added and the plate is incubated at 37 degrees Celsius in a 5% CO2 atmosphere for 15 min. Following this incubation period, 10 ml of rabbit complement (Dynal Biotech Inc., Lake Success, NY) is added to each well. Then, 40 ml (about 4x105 cells/well) of washed, differentiated HL-60 cells are immediately added to each well. The assay plate is incubated at 37 degrees Celsius for 45 min with horizontal shaking (220 rpm). The plate is kept on ice to stop the reaction. A 5 ml aliquot from each well is plated onto an agar medium plate. Plates are incubated overnight at 37 degrees Celsius in a 5% CO2 atmosphere and viable colonies are counted for each well. Typically, 10-60 colonies are expected. The OPK titers will be expressed as the reciprocal of the serum dilution with >/=50% killing compared with the growth in the complement control wells. Serum samples with titers of <8 are reported as a titer of 4 for analysis of the levels of serotype-specific IgG, but excluded for analysis of the correlation between the levels of IgG or HIV-1 viral load and the serum OPK titers. Quality control sera (sera with a known titer) are added to each plate and the blinded test samples for OPK titer are examined only when the titers of quality control sera are identical.

Statistical analyses

All statistical analyses are performed using SAS statistical software (Version 8.1, SAS Institute Inc., Cary, NC, U.S.A.). Categorical variables are compared using 2 or Fisher's exact test whereas non-categorical variables are compared using Wilcoxon's rank-sum test. Univariate analysis followed by multivariate analysis is performed to identify factors associated with 2-fold or greater increase of antibody responses to either one of the three selected serotypes at follow-up for 5 consecutive years. All tests are two-tailed and a p value <0.05 is considered significant.

Implications of the study:

1. If anticapsular IgG response and OPK are significantly higher compare to that of 23-valent pneumococcal vaccination, routine vaccination with 7-valent pneumococcal conjugated vaccine will be suggested for patients with HIV infection.
2. Anticapsular IgG response and OPK will be compared between one dose and two doses groups. Vaccination doses will be suggested according to the results.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients with age >18 years

Exclusion Criteria:

* concurrent immunosuppressant use
* Pregnant women
* receipt of other vaccine within 3 months
* active opportunistic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
2-fold increase of antibody titers specific to pneumococcal serotypes | 48 weeks

SECONDARY OUTCOMES:
antibody titers specific to pneumococcal serotypes larger than 0.35ug/ml All-cause pneumonia | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Ching Hung, MD, MSc, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lu CL, Chang SY, Chuang YC, Liu WC, Su CT, Su YC, Chang SF, Hung CC. Revaccination with 7-valent pneumococcal conjugate vaccine elicits better serologic response than 23-valent pneumococcal polysaccharide vaccine in HIV-infected adult patients who have undergone primary vaccination with 23-valent pneumococcal polysaccharide vaccine in the era of combination antiretroviral therapy. Vaccine. 2014 Feb 19;32(9):1031-5. doi: 10.1016/j.vaccine.2014.01.009. Epub 2014 Jan 15. PMID 24440112